CLINICAL TRIAL: NCT00589082
Title: DaunoXome (Liposomal Daunorubicin) Plus Ara-C Versus Daunorubicin Plus Ara-C in Elderly AML Patients.A Randomized Phase III Study.
Brief Title: DaunoXome + Ara-C vs Daunorubicin + Ara-C in Elderly AML
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Prof. Franco Mandelli, GIMEMA
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GSI 103-AMLE
Record Dates: First submitted 2007-12-24; First posted 2008-01-09 (Estimated); Last update posted 2008-01-09 (Estimated); Status verified 2007-12

CONDITIONS: AML; Elderly
Keywords: AML; elderly; DaunoXome
MeSH Terms: interventions — Daunorubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): standard 3+7
  Interventions: Drug: Daunorubicine
- 2 (Experimental): DNX 3+7
  Interventions: Drug: DaunoXome

INTERVENTIONS:
Drug: DaunoXome
  Arms: 2
Drug: Daunorubicine
  Arms: 1

SUMMARY:
Overall results in the treatment of middle aged adults acute myelogenous leukemia (AML) are substantially improved in the last decade, with complete remission (CR) rates established to values of 70 to 80per cent and also encouraging long-term outcome, especially in patients who can tolerate intensified post remissional treatment strategies. On the contrary, there has been little progress in the treatment of older patients. In these patients the response rate generally range between 40 and 60per cent, and overall survival at 2 years is often less than 10 per cent.

Usually, a combination of anthracyclines daunomycin DNR or doxorubicin and cytarabyne Ara-C has been utilized for the remission-induction treatment, with schedules similar to those utilized in younger cases, for patients eligible to intensive treatments. Variation of the dose of DNR has not brought any significant benefit. The EORTC HOVON randomized trial AML9 compared two drugs in induction for previously untreated patients. DNR versus Mithoxantrone (MTZ). MTZ induction therapy produces a slightly better CR rate than DNR-containing regimen (47per cent vs 38per cent, P equals 0.069), without any significant effect on remission duration and survival. The DFS probability between the two treatment arms was not different. The median DFS estimates were 39 weeks in both groups. The DFS rate at 5 years was 8per cent. Also the duration of survival was similar (p equals 0.23) in the two treatment groups. Median survival estimates were 36 weeks (DNR) and 39 weeks (MTZ). The percentage of patients still alive at 5 years were 6per cent and 9per cent respectively.

DETAILED DESCRIPTION:
It can be stated that single agent DaunoXome seems associated with a level of anti-leukemic activity at least equivalent to the conventional drugs available. In addition, the safety profile of DaunoXome either as a single agent either as a combination with Ara-C seems improved with respect to the conventionally administered anthracyclines. Therefore, it seems warranted to further explore the anti-leukemic activity, the toxicity and the long term results of DaunoXome as a treatment for AML in association with Ara-C against the parent compound daunorubicin. In particular, we propose a study to evaluate standard 3+7 schedule versus the same schedule with DaunoXome instead of daunorubicine as front line treatment in AML patients older than 60 years. Patients achieving a CR will receive a consolidation cycle with the same drugs at the same doses. After consolidation, patients in CR will be randomized to receive a maintenance treatment with low-dose Ara-C plus Atra versus no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Previously untreated AML (including AML after MDS) with > 20% marrow blasts (new WHO classification)
* Age ≥ 61 <75 years
* AML evoluted after MDS are eligible if not previously treated with antiblastic drugs.
* Performance status ≥ 70 (Karnofsky) or ≤ 2 (WHO)
* Signed informed consent from the patient

Exclusion Criteria:

Version 3.0 - february 2001 - CONFIDENTIAL 9

* Patients already treated for their AML with other cytotoxic drugs (except no more than 7 days of Corticosteroids)
* Acute promyelocitic leukemia (FAB M3 or M3v)
* Blast crisis of chronic myeloid leukemia or leukemia supervening after other
* myeloproliferative disease
* Concomitant progressive malignant disease
* Presence of meningeal disease
* History of recent myocardial infarction (within previous 12 months), significant congestive heart failure, life threatening arrhythmia, or cardiovascular disease of Class II or greater according to the New York Heart Association Functional Classification (NYHAFC).
* Abnormal cardiac ejection fraction (45% or less).
* Abnormal hepatic function (ALAT/ASAT or bilirubin >3 N ).
* Abnormal renal function (creatinine >3 N)
* Active bacterial, fungal or viral infection as documented by positive cultures, radiological imaging, clinical signs, septic fever or septic shock symptoms.
* Patients who recover from the infection could be eligible.
* History of hypersensitivity to one of the liposomal constituents.
* Severe pulmonary, neurological or psychiatric disease.
* People unable to give informed consent.
* Presence of any phychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow up schedule.
* HIV positivity
* Intercurrent organ damage or medical problems that would interfere with therapy.

Ages: 61 Years to 75 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-10; Primary Completion 2005-11 (Actual); Study Completion 2005-11 (Actual)

PRIMARY OUTCOMES:
Efficacy and safety of DaunoXome in association with cytosine arabinoside in terms of reduction of induction deaths respect to standard "3+7" chemotherapy

SECONDARY OUTCOMES:
Efficacy, in terms of DFS, of maintenance therapy with low-dose of Ara-C plus ATRA versus no maintenance therapy

CONTACTS AND LOCATIONS:
Overall Officials: Franco MANDELLI, Prof, Principal Investigator — Università di Roma "La Sapienza"

REFERENCES:
- [Background] Zittoun RA, Mandelli F, Willemze R, de Witte T, Labar B, Resegotti L, Leoni F, Damasio E, Visani G, Papa G, et al. Autologous or allogeneic bone marrow transplantation compared with intensive chemotherapy in acute myelogenous leukemia. European Organization for Research and Treatment of Cancer (EORTC) and the Gruppo Italiano Malattie Ematologiche Maligne dell'Adulto (GIMEMA) Leukemia Cooperative Groups. N Engl J Med. 1995 Jan 26;332(4):217-23. doi: 10.1056/NEJM199501263320403. PMID 7808487